CLINICAL TRIAL: NCT03644576
Title: A Phase 1, Randomized, Double-Blind, Placebo-controlled Study to Evaluate the Effect of Ozanimod on Blood Pressure and Heart Rate Response to Pseudoephedrine in Healthy Adult Subjects
Brief Title: Drug-drug Interaction Study of Ozanimod With Pseudoephedrine to Evaluate the Effect on Blood Pressure and Heart Rate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: RPC01-1914; U1111-1215-6267 (Registry Identifier: WHO)
Record Dates: First submitted 2018-08-03; First posted 2018-08-23 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers
Keywords: Ozanimod; Pseudoephedrine; Healthy Adult Subjects
MeSH Terms: interventions — ozanimod; Pseudoephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ozanimod plus Pseudophedrine (Experimental): ozanimod once daily (QD) for 30 days. On Day 30, a single dose of pseudoephedrine 60mg will be co-administered with ozanimod.
  Interventions: Drug: ozanimod; Drug: Pseudoephedrine
- ozanimod placebo plus Pseudoephedrine (Placebo Comparator): ozanimod placebo once daily (QD) for 30 days. On Day 30, a single dose of pseudoephedrine 60mg will be co-administered with ozanimod placebo.
  Interventions: Drug: Pseudoephedrine; Drug: ozanimod placebo

INTERVENTIONS:
Drug: ozanimod — ozanimod
  Arms: ozanimod plus Pseudophedrine
Drug: Pseudoephedrine — Pseudoephedrine
Drug: ozanimod placebo — ozanimod placebo
  Arms: ozanimod placebo plus Pseudoephedrine

SUMMARY:
The purpose of this study is to evaluate the effect of ozanimod after repeated dosing on blood pressure and heart rate response to a single-dose administration of pseudoephedrine (PSE) in healthy adult subjects.

Study Design This is a Phase 1, randomized, double-blind, placebo-controlled study. Approximately sixty eligible subjects will be enrolled and randomized in a 1:1 fashion with 30 subjects in each treatment group.

Subjects will receive placebo or ozanimod once daily (QD) for 30 days. On Day 30, a single oral dose of pseudoephedrine (PSE) 60 mg will be co-administered with placebo or ozanimod.

Study Population The study will enroll approximately 60 healthy men and non-pregnant, non-lactating women, ages 18 to 55 years, inclusive, with a body weight of at least 110 pounds (50 kg) and body mass index within the range of 18.0 to 30.0 kg/m2, inclusive.

Length of Study The study duration is 65 ± 2 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a man or non-pregnant, non-lactating woman, aged 18 to 55 years, inclusive, at the time of signing the informed consent form (ICF).
2. Female subjects must meet at least 1 of the following criteria:

   * Negative serum pregnancy test at Screening and Day -2 (women of child-bearing potential [WOCBP] only).
   * Postmenopausal (defined as 2 years after the last period and follicle-stimulating hormone [FSH] > 40 IU/L).
   * Received surgical sterilization (eg, bilateral tubal ligation, bilateral oophorectomy, hysterectomy) at least 6 months before Screening with medical records.
3. Females of child-bearing potential:

   Must agree to practice a highly effective method of contraception throughout the study until completion of the 75-day Safety Follow-up. Highly effective methods of contraception are those that alone or in combination result in a failure rate of a Pearl index of less than 1% per year when used consistently and correctly.

   Acceptable methods of birth control in this study are the following:
   * Combined hormonal (estrogen and progestogen containing) contraception, which may be oral, intravaginal, or transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation, which may be oral, injectable, implantable
   * Placement of an intrauterine device or intrauterine hormone-releasing system
   * Bilateral tubal occlusion
   * Vasectomized partner
   * Sexual abstinence

   Male subjects:

   Must agree to use a latex condom with spermicide during sexual contact with WOCBP while participating in the study and until completion of the 75-day Safety Follow-up.

   All subjects:

   Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception. Female condom and male condom should not be used together.
4. Male subjects must agree to refrain from donating sperm during the study and until completion of the 75-day Safety Follow-up.
5. Subject has a body weight of at least 110 pounds (50 kg); body mass index (BMI) within the range of 18.0 to 30.0 kg/m2, inclusive, at Screening and Day -2.
6. Subject is in good health, as determined by no clinically significant findings from medical or surgical history, 12-lead ECG, physical examination, clinical laboratory tests, and vital signs.
7. Subject has a mean systolic blood pressure (SBP) of 90 to 140 mmHg, a diastolic blood pressure (DBP) of 50 to 90 mmHg from three consecutive measurements at Screening and Day -2.
8. Subject must be able to comprehend and provide written informed consent, and must be able to comply with the requirements of the study, including the study visit schedule and other protocol requirements

Exclusion Criteria:

1. Subject has clinically significant electrocardiogram (ECG) and cardiovascular symptoms at Screening.
2. Subject has a presence or history of any abnormality or illness that, in the opinion of the investigator, may affect absorption, distribution, metabolism, or elimination of the study drugs or would limit the subject's ability to participate in and complete this clinical study.
3. Subject has a history of clinically significant or unstable vascular disease, or a history of syncope associated with hypotension within the last 2 years or a history of orthostatic hypotension (or SBP decrease of ≥ 20 mmHg 2 minutes after standing compared with supine SBP).
4. Subject with a seated pulse rate outside 55 to 90 beats per minute (bpm) at Screening or Day -2.
5. Subject with a resting Fridericia-corrected interval between Q and T wave in the heart's electrical cycle (QTcF) > 450 msec (males) or > 470 msec (females) or interval from the beginning of the P wave to the beginning of the QRS complex (PR) > 200 msec at Screening.
6. Subject has a history of alcoholism, drug abuse, or addiction within 24 months prior to Screening.
7. Subject has a positive serum test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) at Screening.
8. Subject has used any tobacco- or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, vape, electronic cigarettes, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 3 months prior to the first dose of IP.
9. Subject has consumed any marijuana products within 3 months prior to the first dose of IP.
10. Subject has a positive urine drug test including cotinine at Screening or Day -2.
11. Subject has a positive alcohol urine or breath test at Screening or Day -2.
12. Subject has received any investigational drug within 30 days or 5 times the elimination half-life (if known), whichever is longer, prior to the first dose of IP.
13. Subject has used any systemic over-the-counter medication (excluding acetaminophen up to 1 g/day), dietary or herbal supplement (excluding vitamins/multi-vitamins) within 7 days prior to the first dose of IP. St. John's wort must be discontinued at least 28 days prior to the first dose of IP.
14. Subject has used any systemic prescription medication (excluding hormonal contraceptives) within 28 days or 5 times the elimination half-life, whichever is longer, prior to the first dose of IP.
15. Subject has used any known MAO inhibitors within 90 days prior to the first dose of IP. 16. Subject has a history of allergic reaction to pseudoephedrine or ozanimod.

17. Subject has ingested alcohol within 7 days prior to the first dose of IP. 18. Subject plans or will participate in strenuous physical activities during the 24-hour period prior to the first dose of IP.

19. Subject has poor peripheral venous access. 20. Subject has donated greater than 400 mL of blood within 60 days prior to the first dose of IP.

21. Subject has a history of any medical history that, in the opinion of the investigator, might confound the results of the study or jeopardize the safety or welfare of the subject.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Cardiovascular analysis | Days 29 and 30
  Day 30 maximum time-matched change from Day 29 in systolic blood pressure (SBP)

SECONDARY OUTCOMES:
Pharmacokinetics- Cmax | up to 30 days
  Maximum observed plasma concentration within dosing interval on Days 1, 5, 8, and 28 for ozanimod and its metabolites, and on Day 30 for pseudoephedrine.
Pharmacokinetics- Cmin | up to 30 days
  Minimum observed plasma concentration within the dosing interval
Pharmacokinetics- Tmax | up to 30 days
  Time to Cmax on Days 1, 5, 8, and 28 for ozanimod, and its metabolites, and on Day 30 for pseudoephedrine.
Pharmacokinetics- AUC0-24 | up to 30 days
  Area under the concentration-time curve from time 0 to 24 hours on Days 1, 5, 8, and 28 for ozanimod, its metabolites, total drug and total active drug, and on Day 30 for pseudoephedrine.
Pharmacokinetics- Ctrough | up to 30 days
  Pre- dose or trough concentration for ozanimod and its metabolites on Days 26-30
Adverse events (AEs) | up to 30 days
  Number of participants with adverse events
Pharmacokinetics- % total drug related AUC0-24 for each analyte | up to 30 days
  % total drug related AUC0-24 for ozanimod and each metabolite
Pharmacokinetics- % total active drug related AUC0-24 for each active analyte | up to 30 days
  % total active drug related AUC0-24 for ozanimod and each active metabolite
Cardiovascular analysis for DBP | Days 29 and 30
  Day 30 maximum time-matched change from Day 29 in diastolic blood pressure (DBP)
Cardiovascular analysis for heart rate | Days 29 and 30
  Day 30 maximum time-matched change from Day 29 in heart rate (HR)
Cardiovascular analysis for blood pressure | Days 29 and 30
  Day 30, 24-hour average change from Day 29 24-hour average in Blood pressure (systolic blood pressure (SBP) and diastolic blood pressure (DBP)
Cardiovascular analysis for heart rate | Days 29 and 30
  Day 30, 24-hour average change from Day 29 24-hour average in Heart rate
Cardiovascular analysis for blood pressure | Days 29 and 30
  Day 29 and Day 30 24-hour average for blood pressure (systolic blood pressure (SBP) and diastolic blood pressure (DBP))
Cardiovascular analysis for heart rate | Days 29 and 30
  Day 29 and Day 30 24-hour average for heart rate
Cardiovascular analysis for blood pressure | Days 29 and 30
  Day 30 time-matched changes from Day 29 for blood pressure (systolic blood pressure (SBP) and diastolic blood pressure (DBP))
Cardiovascular analysis for heart rate | Days 29 and 30
  Day 30 time-matched changes from Day 29 for heart rate
Cardiovascular analysis for blood pressure | Days 29 and 30
  Observed blood pressure (systolic blood pressure (SBP) and diastolic blood pressure (DBP))
Cardiovascular analysis for Heart Rate | Days 29 and 30
  Observed heart rate (HR)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Tran, Pharm.D, Study Director — Celgene
Locations (1):
- ICON Early Phase Services, San Antonio, Texas, United States

REFERENCES:
- [Derived] Tran JQ, Zhang P, Walker S, Ghosh A, Syto M, Wang X, Harris S, Palmisano M. Multiple-Dose Pharmacokinetics of Ozanimod and its Major Active Metabolites and the Pharmacodynamic and Pharmacokinetic Interactions with Pseudoephedrine, a Sympathomimetic Agent, in Healthy Subjects. Adv Ther. 2020 Dec;37(12):4944-4958. doi: 10.1007/s12325-020-01500-0. Epub 2020 Oct 6. PMID 33025342